CLINICAL TRIAL: NCT02504593
Title: Novel mHealth Platform to Ensure Quality of Community-based Malaria Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group
Other Study IDs: Pro00063521
Record Dates: First submitted 2015-07-02; First posted 2015-07-22 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Quality Assurance of Malaria Diagnosis
Keywords: Quality Assurance; Monitoring & Evaluation; Malaria rapid diagnostic test (RDT); Community-based malaria diagnosis; Community health workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Community health volunteers (Other): The study subjects are all community health volunteers in community units in Kenya (10 community units in Bungoma East and 6 community units in Kiminini) that have been trained to provide community-based malaria diagnosis through rapid diagnostic testing.
  Interventions: Device: mHealth platform employing Fionet Deki Readers to ensure quality of community-based malaria diagnosis

INTERVENTIONS:
Device: mHealth platform employing Fionet Deki Readers to ensure quality of community-based malaria diagnosis — The investigators propose to implement a new mobile interface that automatically reads and troubleshoots malaria rapid diagnostic test (RDT) cassettes. This device, called a Deki reader (DR), will allow the investigators to establish an extensive quality assurance program of malaria diagnosis performed by trained community health volunteers (CHVs). To ensure high-quality diagnosis by CHVs, the study team will deploy 10 Fionet DRs and rotate them amongst 200 CHVs who have been trained to do RDTs. In the first phase, each CHV will use the device for 10 successive clients presenting themselves for malaria diagnosis to the CHV, and then the device will be rotated to another CHV.

SUMMARY:
The investigators propose to implement a new mobile interface that automatically reads and troubleshoots malaria rapid diagnostic test (RDT) cassettes. This device, called a Deki reader (DR), will allow the investigators to establish an extensive quality assurance program of malaria diagnosis performed by trained community health volunteers (CHVs). The study will lease 10 DRs and rotate them amongst 200 CHVs performing community-based malaria diagnosis through rapid diagnostic testing. The study setting is Bungoma East subcounty and Kiminini subcounty in Kenya. The overall goal is to measure and improve the quality of malaria diagnosis by CHVs using malaria RDTs. The investigators aim for every CHW to exceed 90% sensitivity and specificity and zero operator errors within six months. There are no appreciable risks to the CHV associated with evaluation by the DR device. The investigators' analysis will focus on descriptive statistics of RDT use and accuracy amongst all participating CHVs.

ELIGIBILITY:
Inclusion Criteria:

* All community health volunteers in 10 community units in Bungoma East and 6 community units in Kiminini that have been trained to provide community-based malaria diagnosis through rapid diagnostic testing are eligible.

Exclusion Criteria:

* Any person not meeting the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Percent of RDTs with correct administration and interpretation by CHVs compared across the first and tenth tests | 6 months (during which each consenting CHV of the 200 eligible will conduct 10 tests)
  The percent of RDTs that were properly conducted and interpreted by CHVs, according to Deki Reader results, comparing across the first and tenth RDTs read with the Deki Reader for each CHV.

SECONDARY OUTCOMES:
Percent of RDTs with a false negative reading by CHVs compared across the first and tenth tests | 6 months
  Percent of RDTs with a false negative reading by CHVs compared across the first and tenth tests read with the Deki Reader for each CHV.
Percent of RDTs with a false positive reading by CHVs compared across the first and tenth tests | 6 months
  Percent of RDTs with a false positive reading by CHVs compared across the first and tenth tests read with the Deki Reader for each CHV.
Percent of invalid RDTs not properly identified by CHVs compared across the first and tenth tests | 6 months
  Percent of invalid RDTs not properly identified by CHVs compared across the first and tenth tests read with the Deki Reader for each CHV.
Percent of RDTs that CHVs performed with an improper test procedure compared across the first and tenth tests. | 6 months
  Percent of RDTs that CHVs performed with an improper test procedure compared across the first and tenth tests read with the Deki Reader for each CHV.
Overall sensitivity (measured as the proportion of positive tests as determined by the DR which the CHVs correctly identify). | 6 months
  Overall sensitivity of RDTs performed by CHVs compared to the Deki Reader results. Sensitivity will be measured as the proportion of positive tests as determined by the DR which the CHVs correctly identify.
Overall specificity (measured as the proportion of negative tests as determined by the DR which the CHVs correctly identify). | 6 months
  Overall specificity of RDTs performed by CHVs compared to the Deki Reader results. Specificity will be measured as the proportion of negative tests as determined by the DR which the CHVs correctly identify.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy O'Meara, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Eldoret, Kenya